CLINICAL TRIAL: NCT00787956
Title: Evaluation of an Internet Chronic Disease Self-Management Program for Australia
Brief Title: Internet Chronic Disease Self-Management Program for Australia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kate Lorig, professor emertius, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SU-10032008-1315
Record Dates: First submitted 2008-11-06; First posted 2008-11-10 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

INTERVENTIONS:
Behavioral: Internet Chronic Disease Self-Management Program (ICDSMP)

SUMMARY:
The Internet Chronic Disease Self-Management Program (ICDSMP) is a pilot study of our existing, previous approved, Chronic Disease Self-Management Program Online. The online programme will be offered to 300 people with chronic disease in South Australia and evaluated for effectiveness, as well as satisfaction of both the South Australian peer facilitators and the participants with chronic disease. All participants will be recruited by the State of South Australia, after which they will complete informed consent and a questionnaire on a secure website housed at Stanford. They will take a 6-week online self-management program in groups of 20-25, and they fill our additional online questionnaires at 6 month and one year.

DETAILED DESCRIPTION:
The study will determine if the ICDSMP can be effective in the diverse population of South Australia. We hope that this online workshop will provide South Australians easy access to the Chronic Disease Self-Management Workshop. If successful, this program or similar programs could be made broadly available. The workshop being offered on the internet will offer this program as an alternative mode of service delivery to support self-management education for chronic diseases and will become an integral part of high quality primary health care in the state.

1. A potential subject will learn of the project through advertisement done by existing community CDSMP providers or by websites or online newsletter provided by State of South Australia. The announcements will direct them to the study website at Stanford, where they will read a description of the project and leave their names and email addresses if they are interested in participating.
2. When enough people are on the wait list to fill an online workshop, Stanford will send an email with a unique URL for each potential participant to log on, complete the informed consent, and fill out the baseline questionnaire. They will create their own username and password during this process.
3. Once 24 people have enrolled, they will be assigned to a workshop and receive an email detailing when the workshop starts and inviting them to log on to familiarize themselves with the online environment and meet their moderators and other classmates online.
4. They will start the 6-week workshop with each session starting a week apart with new content. They are expected to log on 2-3 times per week, for a total time of about 2 hours. They may log on more often if they wish, and they are not required to log on at any specific time.
5. The workshop consists of didactic/interactive web pages, 4 discussion boards, an internal anonymous message center, a section of personalized tools that are available only to the individual participant and Stanford staff, and a help section. Each workshop is facilitated by 2 trained peer moderators, supervised by Stanford staff.
6. The moderators offer help to those who may be confused by the goal setting exercise, for example, to give feedback to participants' progress, and to remind people to log on if they have not. They monitor for safety.
7. After the end of the 6-week workshop, participants will be able to log into the workshop to review the past 6-weeks' participation and print out any useful workshop materials for future reference
8. 6 months after the end of the 6-week workshop, participants will complete a follow up questionnaire, and again at 1 year.

ELIGIBILITY:
Inclusion Criteria:- be 18 or older

* live in South Australia
* have at least one long term condition (It is suitable for people with heart disease, lung disease, or type 2 diabetes as well as other diagnosed chronic condition)
* and be able to fill out the on-line questionnaire without assistance.
* Have access to the internet and an email account
* Able to read English Exclusion Criteria:be pregnant
* if they self-identify they are enrolled in another program similar to this one, they will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Health Status | 6 an 12 months

SECONDARY OUTCOMES:
Health behaviors | 6 and 2 months
Health care utilization | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kate R Lorig, Principal Investigator — Stanford University
Locations (2):
- Stanford University School of Medicine, Stanford, California, United States
- Country Health SA, Mount Gambier, South Australia, Australia